Date: 14-07-2023

Protocol version 01.01.03

# Fibrosis, inflammation, Oxygenation of Renal Tissue In FabrY disease: The FORTIFY study

#### Project group

- Caroline Kistorp<sup>1</sup>, professor, MD, PhD
- Niels H. Brandt-Jacobsen<sup>1, 2</sup>, MD, PhD-studerende
- Ulrik B. Andersen<sup>2,3</sup>, MD, PhD
- Bryan Haddock<sup>2,3</sup>, BSc, PhD
- Henrik Larsson<sup>2,3</sup>, professor, MD, PhD

#### Institution

<sup>1</sup>Department of Hormone and Metabolism, Centre of Cancer and Organ Diseases, University Hospital of Copenhagen - Rigshospitalet, Copenhagen, Denmark

<sup>2</sup>Department of Clinical Physiology and Nuclear Medicine, Centre of Diagnostics, University Hospital of Copenhagen – Rigshospitalet, Copenhagen, Denmark

<sup>3</sup>The Functionel Imaging Unit, Centre of Diagnostics, University Hospital of Copenhagen – Rigshospitalet, Copenhagen, Denmark

### Sponsor, initiator, and principal investigator

Caroline M. Kistorp, MD, PhD, Professor,
Department of Hormone and Metabolism,
Centre of Cancer and Organ Disease,
University Hospital of Copenhagen – Rigshospitalet
Blegdamsvej 9
DK-2100 Copenhagen, Denmark

Telephone: +45 22 47 56 99 / +45 35 45 96 42 Email: caroline.micheala.kistorp@regionh.dk

#### Specialist registrar

Niels Høeg Brandt-Jacobsen, MD, Ph.D, Post.doc

Date: 29-08-2023

Protocol version: 01.01.3

Overreaching aim

The overall objective of this study is to investigate Fabry-associated renal organ involvement by

using a novel magnetic resonance imaging (MRI) approach, focusing on changes in renal oxygen

levels by blood oxygenation-level dependent (BOLD) imaging. Furthermore, to correlate renal

oxygenation to the phenotypic presentation of patients with Fabry-associated nephropathy regarding

circulating and imaging-derived biomarkers of kidney inflammation, fibrosis and injury as

compared with healthy age- and sex-matched controls.

The study will achieve this by:

1) Using a non-invasive, contrast-free MRI protocol focusing on parameters of oxygenation,

inflammation, fibrosis, and injury in the kidney.

2) Using an extensive, in-depth biomarker blood panel to investigate the pathological pathways

associated with Fabry disease and Fabry-associated nephropathy.

Introduction

Fabry disease is a rare X-linked lysosomal disorder caused by mutations in the gene encoding the

enzyme  $\alpha$ -galA, an essential enzyme for normal cellular function. The enzyme deficiency causes

progressive accumulation of glycosphingolipids, especially globotriaosylceramide (Gb3) in virtually

all organs, leading to dysfunction and eventually leading to organ failure. Although, Fabry disease

is caused by an X-linked genetic mutation and the clinical implication among men with a classic

phenotype are most severe, Fabry disease affects both males and females [1]. Men with a non-classic

phenotype and females present with a more heterogenous degree of organ involvement, however,

these patients remain at increased risk of multisystem organ involvement and must be attend

extensive screening, evaluated repeatedly in order to decide when and who are in need of treatment

[2]. However, as evident in patients with the several known genotypes, which presents with no or

very low  $\alpha$ -galA-activity and develop early multi-organ involvement, one of the complication of

greatest prognostic impact is an early involvement of the kidney [1].

Fabry nephropathy

Although, the etiology of kidney affection in Fabry disease in general is well established, the actual

mechanisms of progression – and thus the targets of therapeutic approach – are largely unknown.

Fabry nephropathy is characterized by the accumulation of Gb3 deposition in podocytes, epithelial

cells and endothelial cells throughout the tubules, where kidney biopsies suggest healthy,

functioning tissue is substituted with reparative diffuse fibrosis. Indeed, evidence shows a direct


Date: 29-08-2023

Protocol version: 01.01.3

association between Gb3 accumulation and both a decline in renal glomerular filtration rate and an increase in urinary albumin excretion – both clinically validated biomarkers of kidney injury and decline in function [3–5]. Given Gb3 accumulation in Fabry disease accounts for less than 5% of the total tissue volume at maximum [6,7], the disproportionate and devastating effects observed have led to the proposal of Gb3 having additional effects beyond mere storage [8–11]. Oxidative stress, endothelial dysfunction, and inflammation have been proposed as important mechanisms induced directly or indirectly by Gb3 accumulation, resulting in increased cell-death of functioning glomeruli with unamenable, reparative fibrosis as a result [9–12]. Furthermore, certain cells seems more susceptible to injury and less susceptible to the benefits expected from Fabry-specific treatment; an important example being renal podocytes [3].

#### Fabry nephropathy and Magnetic Resonance Imaging

Renal hypoxia is now considered to play a key role in the development of chronic kidney disease (CKD) [13–17]. Using a novel contrast-free, non-invasive magnetic resonance imaging (MRI) [16], our collaborative partners have reported renal hypoxia in subjects with type I diabetes and pathological urinary albumin/creatinine ratio (UACR) levels [18]. Recent advances in MRI thus, enables us to investigate the pathological mechanisms underlining Fabry nephropathy by noninvasively measurements of oxygenation, inflammation and fibrosis [13-16]. The kidney's oxidative capacity evaluated by R2\*-related blood oxygenation level-dependent (BOLD) MRI has been validated as a parameter of renal cortical and medullar oxygen-partial pressure [13–16]. Furthermore, changes in dynamic R2\*-signaling have been validated as a non-invasive, contrastfree measure of renal oxygenation capacity, which becomes reduced with presence of chronic kidney disease [14,16]. Concurrently, arterial spin labelling (ASL) is able to provide a reliable measure of total blood flow as well as regional blood flow in the renal artery and the kidney [14,16]. Finally, the inflammatory and fibrotic burden can be elucidated upon by diffusion-weighted sequences and native T1-mapping [13,16]. Therefore, this novel method provides information on kidney-specific shift in energetic oxygen-dependent capacity, ongoing inflammation, and accumulation of fibrosis, with changes not only portraying key aspects of kidney physiology, but changes expected to elucidate on the pathophysiology forming the very basis of Fabry nephropathy.

While the recent advances in imaging present a unique possibility for early detection of Fabry nephropathy, there is a need for validation against clinically established biomarkers of risk such as pathologically increased UACR – currently the greatest predictor of progressive loss of glomerular function in regards to end-stage renal disease in general and in Fabry nephropathy [4,5]. Pathological UACR levels is considered the first clinical sign of Fabry nephropathy, with an estimated prevalence

Date: 29-08-2023

Protocol version: 01.01.3

of 50% among men aged 35 years. Even among women, which often less severely afflicted, up to

40% develop proteinuria and 15% experience a clinically significant renal event, thus, the prognostic

importance of increased UACR in Fabry disease is evident [19-21]. Therefore, UACR levels is the

key clinical parameter of Fabry nephropathy as recommended in guidelines [22].

**Hypothesis** 

Impaired renal oxygenation is an early characteristic of Fabry nephropathy, which precedes

established markers of renal decline such as estimated glomerular filtration rate or UACR.

Participants and methods

Study design

A cross-sectional study and will consist of a group of patients from the Danish National Fabry

Cohort followed at the Danish National Fabry Centre, Department of Hormone and Metabolism,

Copenhagen University Hospital, Rigshospitalet. Furthermore, a control group of healthy age- and

sex-matched individuals will be included to comprise a contemporary control cohort and will

undergo the same program.

**Participants** 

We will enroll 40 participants with Fabry disease previously verified by genetic testing. The Fabry

patients will be divided into two groups with and without renal involvement. Renal involvement is

defined according to UACR levels and impairment of kidney function using the KDIGO

classification [23].

• n=20: UACR  $\ge$  30 mg/g and eGFR < 60 ml/min/1.73m<sup>2</sup> ( $\ge$  CKD G3a/A2).

• n=20: UACR < 30 mg/g and eGFR  $\geq$  60 will be included ( $\leq$  CKD G2/A1).

A control group will consist of 20 healthy age- and sex-matched controls with no renal impairment

( $\leq$  CKD G2/A1: UACR < 30 mg/g and eGFR  $\geq$  60 ml /min).

Inclusion and exclusion criteria

Fabry cohort

**Inclusion criteria** 

- Male and female individuals with a genetically-verified diagnosis of Fabry disease

-  $\geq$  18 years of age.


Date: 29-08-2023

Protocol version: 01.01.3

- Able to give informed consent

#### **Exclusion criteria**

 Any contraindication for magnetic resonance imaging according to standard checklist used in clinical routine, including claustrophobia or metallic foreign bodies, metallic implants, internal electrical devices, or permanent makeup/tattoos that cannot be declared MR compatible.

- Pregnancy

#### Control group

#### **Inclusion criteria**

- Male and female individuals (≥18 years of age)
- Able to give informed consent

#### **Exclusion criteria**

- A genetically-verified diagnosis of Fabry disease.
- Family member to a patient with a genetically-verified diagnosis of Fabry disease
- Cancer expected to influence life expectancy.
- Known heart failure, previous apoplexia or previously established kidney disease.
- Initiation or change of antihypertensive therapy within 3 months of enrolment
- Renal impairment as depicted by the CKD-EPI classification (≥ CKD G2/A1)
- Any contraindication for MRI according to standard checklist used in clinical routine, including claustrophobia or metallic foreign bodies, metallic implants, internal electrical devices, or permanent makeup/tattoos that cannot be declared MR compatible.
- Pregnancy

# **Endpoints**

#### Primary endpoint

A between-group difference in renal hypoxia (R\*) evaluated by BOLD MRI when comparing the groups of patients with Fabry disease.

#### Secondary endpoints

- A between-group difference in renal hypoxia (R\*) evaluated by BOLD MRI when comparing patients with Fabry disease irrespective of renal impairment with the control group.

Date: 29-08-2023

Protocol version: 01.01.3

- A between-group difference in perfusion of the renal cortex (mL/100g/min) when comparing patients with Fabry disease with the control group.

- A between-group difference in perfusion of the renal medulla (mL/100g/min) when comparing groups with Fabry disease patients with the control group.
- A between-group difference in renal blood flow (mL/min) when comparing groups with Fabry disease patients with the control group.
- A between-group difference in native T1 (ms) when comparing groups with Fabry disease patients with the control group.
- A between-group difference in diffusion-weighted signaling when comparing groups with Fabry disease patients with the control group.

#### **Procedures**

#### **Imaging procedure**

MRI scanning of renal hemodynamics and oxygenation

The scanning protocol will consist of one scanning session (hereafter *RENOXY* scan) (Table 4). In brief, the RENOXY scan will consist of sequences of oxygenation (R2\*-BOLD), perfusion (ASL), renal arterial flow (phase contrast), inflammation (T1), fibrosis (diffusion-weighted), preceded by a structural mapping sequence. In addition, a shorter version will be repeated during inhalation of 100% oxygen, including only structural mapping, BOLD, ASL and phase-contrast.

The entire session will last approximately 40-45 minutes (Table 1). If a participant is unable to endure the full scanning protocol a shortened version can be used. All scans will be performed on the same 3-T Philips Achieva.

| Table 1: RENOXY scan | | |
|---|---|---|
| Procedures | Sequences | Time (app.) |
| Rest | 30 minutes of rest prior to scanning sequence | |
| MRI session | - RENOXY scan | 35 min |
| | - Hyperoxygenation scan | 10 min |

#### Clinical procedures

In addition to the imaging protocol, the participants will receive a full clinical work-up, fill out questionnaires in addition to blood and urine-sampling (Table 2).

Date: 29-08-2023 Protocol version: 01.01.3

| Table 2: Clinical procedures | |
|---|---|
| Procedures | Outcome |
| Semi-structured interview | - Medical history, including concomitant chronic disease, |
| | current medication, and dietary supplements. |
| | - Alcohol, tobacco, and substance abuse |
| | - Socioeconomic status and educational background |
| Clinical examination | - Anthropomorphic measures (Age, height, weight, waist and hip |
| | circumference, body mass index [BMI, kg/m <sup>2</sup> ]) |
| | - Office blood pressure and pulse |
| | - Electrocardiogram |
| | - Examination as specified in the |
| | - Mainz Severity Score Index |
| | - Fabry international prognostic index |
| Patient reported outcome | - "Dit helbred og velbefindende" (SF-36®; Quality of life) |
| | - |
| Blood and urine samples | Research Biobank focusing on |
| | - Kidney function, inflammation, and fibrosis and cellular |
| | signaling in the kidney |
| | - Metabolic dysfunction |
| | - Risk markers of disease |
| | - Markers related to Fabry disease risk and progression |
| | Establishing a biobank of future research |
| | - Surplus biological material acquired will be kept in a biobank |
| | for future research. |
| | See table 3 for overview of biomarkers |

#### Medical interview and clinical examination.

Participants will undergo a semi-structured interview to acquire relevant patient information such as, but no limited, to their previous medical history, established concomitant disease, current medication, their use of dietary supplements, their use of alcohol, tobacco and substance abuse, their socioeconomic, and educational background.

They will undergo a focused clinical examination acquiring basic anthropomorphic measures such as age, height, weight, hip- and waist circumference. Furthermore, the clinical examination will

Date: 29-08-2023

Protocol version: 01.01.3

consist of general health measures such as office blood pressure, pulse, electrocardiogram, and a physical examination specified to fulfill the elements of a modified Mainz Severity Score Index and the Fabry International Prognostic Index.

#### Patient reported outcome

Participants will be asked to answer health-related questionnaires and questionnaires regarding their current symptoms and their severity. These questionnaires are used and validated in Fabry disease and include:

- The SF36 Quality of Life-questionnaire

#### Blood and urine sampling

Participants will be required to undergo standard antecubital venipuncture to sample blood. The amount drawn will be 300 mL at the study visit. Regarding urine sampling, participants are to provide a first-voided, morning urine sample.

All samples, which are kept in the research biobank, are acquired and immediately frozen as aliquots and subsequently stored at -80 degrees (Celsius) until the end of the trial. The research biobank is to cease 6 months after last patient last visit; scheduled at 01.12.2025. At the day the research biobank ceases, the remaining material will be considered surplus and will be transferred to the biobank of future research. Regarding the research biobank, when performing the planned analysis, samples are to be thawed and analyzed in immediate succession, with repeat intra- and inter-assay analyses to determine and validate analysis-specific variation according to local laboratory standards. Postponing analysis until end of study is done to minimize time-dependent variation and is deemed necessary as part of trial conduct. Surplus material – both blood and urine – is stored and kept, comprising a biobank of future research. The biobank of future research is established and kept in accordance with the Danish laws on Data Protection and Data Security.

Biomarkers of interest to be analyzed on samples of blood or urine are specifically defined in protocol (table 3). Although all biomarkers are chosen due their prospective or established clinical value, further biomarkers may be necessary to be defined at a later date (e.g. omcis-based blood or urinary biomarker panel). If one or more biomarkers of interest are thought of post-hoc, a new informed consent is required. However, a relevant ethical committee can provide dispensation regarding renewed consent. Separate consent forms will be signed in regard to the research biobank and the biobank of future research, respectively (SeeConsent forms).

Date: 29-08-2023 Protocol version: 01.01.3

| Table 3: Pre-specified biomarkers in research biobank | | |
|---|---|---|
| Sample | Biomarker | Volume |
| Blood | <ul> <li>Circulating biomarkers specific to Fabry's Disease</li> <li>α-gal A activity in leucocytes, Lyso-Gb3 and Gb3, and urine Gb3 Kidney function, fibrosis and inflammation, and cellular signaling in the kidney</li> <li>Creatinine, GDF-15, TGF-β, FGF-21, and FGF-23, VEGF, collagens</li> <li>Clinical biomarkers of metabolic dysfunction</li> <li>fasting plasma glucose, insulin, 3-OH-hydroxybutyrate, HbA1c, and lipid profile.</li> <li>Biomarkers of cardiorenal risk</li> <li>NT-proBNP, TnI, hsTnT, proANP, proCNP</li> </ul> | 300 mL |
| Urine | Urinary excretion - urinary podocyte excretion, ACR | 200 mL |

#### Study visits

Participants eligible for inclusion in the study will be required to attend 1 study visit to participate in the study program. However, if the participant is unable to attend a full study visit at any one day, the scanning protocol can be performed on a separate day from the remaining procedures.

## Statistical considerations

# Justification of sample size

From our previous study, we found that the mean baseline R2\* was 23 with (SD=4). A between-group difference in R2\* of 2.0 units can be considered a clinically important difference [24]. In the cohort, a difference of 2.0 units, an SD of the difference of 2, 80% power, a type 1 error of 5%, and wanting to compare groups independently results in a need of randomizing 51 participants 1:1:1 – corresponding to 17 participants in each group. Accounting for incident claustrophobia causing an unexpected loss of data, we aim to include 20:20:20 participants (Fabry w/ renal impairment; Fabry w/o renal impairment; age- and sex-matched controls).

The current study is an observational cross-sectional study, and the power calculation is performed to investigate the relationship between the presence of renal impairment with the phenotypic presentation of Fabry nephropathy. As the current Danish National consists of 100 individuals, of which approximately 40% have a history albuminuria, a study size consisting of 40 patients with genitically-verified Fabry disease will be feasible in the current patient population.

Furthermore, a simultaneously included control cohort of 20 healthy age- and sex-matched control, will constitute a basis for an in-depth comparison on the clinical implication of biomarkers

Date: 29-08-2023

Protocol version: 01.01.3

not readily available as part of routine clinical screening and is considered necessary as part of study

conduct.

Risks and discomforts

There can be unexpected risks and discomforts attributable to participation in the study, which

cannot be predicted prior to trial conduct. The following will elaborate on known risks and

discomforts.

Risks related to clinical procedures

**Blood sampling** 

Venipuncture to acquire blood samples can be uncomfortable but is considered safe and performed

as a routine procedure in standard medical practice. Although a small hematoma may occur, and a

minimal risk of infection is present, proper technique will be applied to ensure a minimal level of

risks. In comparison to blood donation, where 500 mL is drawn, the current study will require a

sample of 300 mL and may induce slight, transient lightheadedness, but is otherwise not associated

with any known risk.

Additional risks related to scanning procedures

Magnetic resonance imaging

MRI is considered safe and is not related to short- or long-term risk. If a participant becomes

claustrophobic and wants to terminate an ongoing exam, the physician is obliged to do so. In relation

to the scanning procedure, participants are required to breathe while inhaling 100% oxygen during

imaging. This procedure is not associated with any known short-term or long-term risks or

discomforts.

Studies have shown fetus heart rate increases while performing MRI scans. This change is

interpreted as a sign of fetal stress, why pregnancy is a contraindication to trial participation.

Data protection of Personal Information in the Study

All legislations, regulations, and laws on Data Protection and Data Security and the directives of the

Danish Protection Agency will be complied with during the conduct of the trial. Permission to handle

personal data will be sought and approved by the Danish Data Protection Agency. All data are stored

pseudo-anonymized and analyzed electronically and no unauthorized access to data is allowed.


Date: 29-08-2023

Protocol version: 01.01.3

Original data is filed according to a unique participant number. REDCap, hosted by OPEN (Open Patient data Explorative Network) will be used for registration of clinical data. REDCap meets the safety requirements set by the Danish Data Protection Agency for storage of person-sensitive data; prescribed medication, medical history, height, weight are examples of such data. Data will be encrypted and stored for 15 years in accordance with recommendations on data storage from the Danish Data Protection Agency and thereafter transferred to the Danish Data Archives.

The study is reported to the Danish Data Protection Agency in Region H and will be handled according to the regulations of the General Data Protection Regulation: GDPR: REGULATION (EU) 2016/679 OF THE EUROPEAN PARLIAMENT AND OF THE COUNCIL of 27th of April 2016 on the protection of natural persons with regard to the processing of personal data and on the free movement of such data, and repealing Directive 95/46/EC and the Act on Processing of Personal Data. Data is stored for 15 years.

# Procedures for recruiting participants and informed consent

#### **Initial contact**

Fabry patients are recruited from the Department of Hormone and Metabolism, Copenhagen University Hospital, Rigshospialet. The department is assigned as the national center concerning the treatment and monitoring of patients with Fabry disease. Eligibility to participate is evaluated by the doctor or other personnel of the patient's usual care at a regularly scheduled outpatient visit. Eligibility is evaluated using a confirmed diagnosis of Fabry disease using the current clinical standard, UACR and eGFR, and these three parameters (i.e. the inclusion criteria) will be transferred to the project doctor - UACR and eGFR are key parameters of renal function for the inclusion to the project. Patients who fulfill the inclusion criteria and none of the exclusion criteria will be informed of the study by the personnel at the department involved in their usual care. By acceptance, they will receive a written patient information. If the patient favors contact initiated by an investigator from the study and provides oral consent, the patients contact information (name, email, phone number) will be forwarded to an investigator. The oral information for the study is then presented by a medical doctor, who is a member of the study group at the department, given in quiet surroundings. Individuals acting as controls in the study will be recruited from varies homepages (sundhed.dk, facebook, and forsoegspersonen.dk), where contact information on investigators can be found. The recruitment material will be reviewed and approved by the Ethics Committee prior to use. Potential participants can contact the Departments of Hormone and Metabolism, Copenhagen University Hospital, Rigshospitalet by email or telephone. Regarding advertisements on Facebook,

Date: 29-08-2023

Protocol version: 01.01.3

any advertisement/post will have its ability to be shared or write a comment to the advertisement/post disabled. In addition to the written information pertaining to the study, it will be accompanied by the brochure: "Forsøgspersoners rettigheder i et sundhedsvidenskabeligt forskningsprojekt" (Your rights as a participant in medical research) and "Dit væv, din ret" (Your tissue, your right). If the individual accepts further information on the study, a meeting in a quiet, undisturbed room will be scheduled with one of the investigators, and the person will be informed of the right to have a bystander present at that moment. The patient will be offered at least 24 hours reflection period before signing the consent form. The informed consent to participate in the study gives the research responsible doctors, sponsor and their representatives, and potential control authorities access to the information on kidney function, and relevant medical information for the study from the patient's medical record.

**Scheduled meeting** 

At the scheduled meeting, the individual will receive additional oral information, from an investigator, and it will be clarified whether the patient fulfill the general participation criteria. The patient will be informed about the terms and restrictions of the form of 'informed written consent'. The investigator will ensure that the patient is adequately informed about the study background and design both orally and in writing. It will be made clear that the patient can withdraw from the study at any time without repercussions.

Acquisition of informed consent

If the patient is interested in participating in the study after the initial information meeting and after the allotted deciding time, a meeting will be scheduled where oral and written informed consent will be obtained. After consent to participate in the study has been obtained, the first study visit will be scheduled. No study-related examinations will be conducted prior the acquisition of informed consent. Investigators will only access electronic hospital records to transfer or record information after acquisition of written informed consent.

**Informed consent** 

The participant will be required to sign the individual forms of informed consent applicable.

Consent regarding study participation

The participant's consent includes the right to read and transfer information from electronical hospital records to RED-Cap by investigators. The data transferred include information such as medical history, blood and urine test results, prescribed and over-the-counter medication. Further,

Date: 29-08-2023

Protocol version: 01.01.3

the informed consent includes permission to establish a research biobank regarding the analyses of biomarkers specified in the protocol. In addition, consent gives direct access to electronic hospital records for the primary investigator, the sponsor or their representatives, as well as authorized auditors in order to retrieve the health-related information necessary to perform the study and to perform quality control and monitoring. The access to electronic hospital records gives access to information from previous clinical evaluations performed by doctors or other hospital staff in relation to hospitalizations or outpatient visits as well as previously performed diagnostic analysis (e.g. biochemical analysis of blood, urine or other tissue samples), image-based evaluations (e.g. by ultrasound, computer-tomography or magnetic resonance imaging), and previous and current use of prescribed medication. These sources of information are vital in order to acquire a sufficient image of the patient's current medical health status.

The informed consent will be valid for the duration of the study.

#### Consent regarding establishment of a biobank of future research

A separate form of informed consent gives permission of the establishment of a biobank of future research consisting of extra material, if any, acquired at the initial visit of the core program. The aim of the biobank for future research is to ensure the ability to answer contemporary research questions in a rapidly evolving field. Future analyses may therefore include, but not be limited to analyses of circulating levels of hormones, proteins, DNA-excerpts, not specified in the current protocol. Future analyses will be required to be approved by the regional ethics committee prior to analysis.

The informed consent will be valid for the duration of the study.

#### Time schedule

| - | Ethics committee approval | 01.08.2023 |
|---|------------------------------------------------|------------|
| - | First patient first visit | Q4, 2023 |
| - | Last patient last visit | Q2, 2025 |
| - | Cessation of Research Biobank | 01.12.2025 |
| - | End of data analysis and manuscript submission | Q4, 2025 |

Data acquired is stored for 15 years after acquisition. The biobank of future research is created at the date of cessation of the research biobank.

## **Funding**

The study will be funded by external independent private and public foundations. Any funding is deposited in a research account administered at Rigshospitalet, Copenhagen University Hospital -

Date: 29-08-2023

Protocol version: 01.01.3

Rigshospitalet, Denmark. None of the investigators or departments will have any financial gain from conducting the study. As funding is secured, the ethical committee (VEK) and the included patients will be informed, and the patient information will be accordingly updated to include the information on funding sources.

#### Patient insurance and reimbursement

The study is conducted at the Department of Hormone and Metabolism, Rigshospitalet and covered by the departments insurance. Participants in the trial are covered by the existing patient insurance ("Patienterstatningen"). The participants will not receive payment. If the study requires extra visits to the department, transportation cost will be covered according to the guidelines for voluntary research subject's appendix 1 of the National Scientific Committee (NVK). Furthermore, expenses as to their nutritional need during visits will be provided for.

# Ethical considerations and clinical implications

The study will be conducted in accordance with the Helsinki II declaration, the regulations of the General Data Protection Regulation, and will follow the directives of the laws on Data Security ('Datasikkerhed') and on Data Protection ('Databeskyttelsesloven'). The study will be approved by the Danish Data Protection Agency and the Regional Ethics Committee of Copenhagen Denmark. Furthermore, the trial will be conducted following the current clinical research standard. The study is to undergo independent monitoring ensuring trial conduct in accordance with the guidelines of Good Clinical Practice (GCP). By following GCP, it is ensured that the data collected is valid, complete, and well-documented. Anonymity of the participants is explicitly guaranteed.

Kidney disease is one of the complications with the greatest clinical impact in Fabry disease. Using a cutting-edge MRI-based approach, we will uncover and broaden the understanding of renal pathophysiology and its involvement in Fabry disease. All scheduled procedures, with the exception of the MRI scan, are a part of the current clinical observational program for patients with Fabry Disease at the Danish National Fabry Center. The addition of magnetic resonance imaging of the kidneys – the main focus of this trial – is considered a safe procedure and carries no additional risk. We believe the planned program will provide evidence of incremental value in a rare genetic disease associated with impairment of multiple organ systems, which progress faster, and leads to organ failure at an earlier age than seen in the general population. Therefore, we believe the current study will improve the diagnostic approach and the ability to detect patient in early stages of disease. Furthermore, we find that the potential therapeutic gain for the participants and future patients

Date: 29-08-2023

Protocol version: 01.01.3

outweigh the risks and discomforts of participating in the study, and therefore, we believe

conducting the study is justified.

Dissemination of results

The investigators oblige themselves to publish all clinically relevant findings in peer-reviewed

journals irrespective of their ability to achieve statistical significance – i.e. publishing all results

irrespective of being positive, neutral, or negative. Results will be published following the

International Committee of Medical Journal Editors (ICMJE) recommendations.

The investigators will present findings at national and international conferences with an aim to

strengthen the current understanding of, to substantiate or challenge the current clinical approach to

Fabry disease. Furthermore, the authors will disseminate the results of the overreaching aims among

patients with Fabry disease through patient organizations on the national level.

Date: 29-08-2023 Protocol version: 01.01.3

# References

- [1] Waldek S, Patel MR, Banikazemi M, Lemay R, Lee P. Life expectancy and cause of death in males and females with Fabry disease: Findings from the Fabry Registry. Genet Med 2009;11:790–6. https://doi.org/10.1097/GIM.0b013e3181bb05bb.
- [2] Wanner C, Germain DP, Hilz MJ, Spada M, Falissard B, Elliott PM. Therapeutic goals in Fabry disease: Recommendations of a European expert panel, based on current clinical evidence with enzyme replacement therapy. Mol Genet Metab 2019;126:210–1. https://doi.org/10.1016/j.ymgme.2018.04.004.
- [3] Najafian B, Tøndel C, Svarstad E, Gubler MC, Oliveira JP, Mauer M. Accumulation of globotriaosylceramide in podocytes in fabry nephropathy is associated with progressive podocyte loss. J Am Soc Nephrol 2020;31:865–75. https://doi.org/10.1681/ASN.2019050497.
- [4] Germain DP, Hughes DA, Nicholls K, Bichet DG, Giugliani R, Wilcox WR, et al. Treatment of Fabry's Disease with the Pharmacologic Chaperone Migalastat. N Engl J Med 2016;375:545–55. https://doi.org/10.1056/nejmoa1510198.
- [5] Jehn U, Bayraktar S, Pollmann S, Van Marck V, Weide T, Pavenstädt H, et al. α-Galactosidase a Deficiency in Fabry Disease Leads to Extensive Dysregulated Cellular Signaling Pathways in Human Podocytes. Int J Mol Sci 2021;22. https://doi.org/10.3390/ijms222111339.
- [6] Linhart A, Elliott PM. The heart in Anderson-Fabry disease and other lysosomal storage disorders. Heart 2007;93:528–35. https://doi.org/10.1136/hrt.2005.063818.
- [7] Yogasundaram H, Kim D, Oudit O, Thompson RB, Weidemann F, Oudit GY. Clinical Features, Diagnosis, and Management of Patients With Anderson-Fabry Cardiomyopathy. Can J Cardiol 2017;33:883–97. https://doi.org/10.1016/j.cjca.2017.04.015.
- [8] Eikrem Ø, Skrunes R, Tøndel C, Leh S, Houge G, Svarstad E, et al. Pathomechanisms of renal Fabry disease. Cell Tissue Res 2017;369:53–62. https://doi.org/10.1007/s00441-017-2609-9.
- [9] Ravarotto V, Simioni F, Carraro G, Bertoldi G, Pagnin E, Calò LA. Oxidative stress and cardiovascular-renal damage in fabry disease: Is there room for a pathophysiological involvement? J Clin Med 2018;7:1–7. https://doi.org/10.3390/jcm7110409.
- [10] Sanchez-Niño MD, Carpio D, Sanz AB, Ruiz-Ortega M, Mezzano S, Ortiz A. Lyso-Gb3 activates Notch1 in human podocytes. Hum Mol Genet 2015;24:5720–32. https://doi.org/10.1093/hmg/ddv291.
- [11] Ravarotto V, Carraro G, Pagnin E, Bertoldi G, Simioni F, Maiolino G, et al. Oxidative stress and the altered reaction to it in Fabry disease: A possible target for cardiovascular-renal remodeling? PLoS One 2018;13:1–14. https://doi.org/10.1371/journal.pone.0204618.
- [12] Fall B, Scott CR, Mauer M, Shankland S, Pippin J, Jefferson JA, et al. Urinary podocyte loss is increased in patients with fabry disease and correlates with clinical severity of fabry nephropathy. PLoS One 2016;11:1–14. https://doi.org/10.1371/journal.pone.0168346.
- [13] Selby NM, Blankestijn PJ, Boor P, Combe C, Eckardt KU, Eikefjord E, et al. Magnetic resonance imaging biomarkers for chronic kidney disease: a position paper from the European Cooperation in Science and Technology Action PARENCHIMA. Nephrol Dial Transplant 2018;33:ii4–14. https://doi.org/10.1093/ndt/gfy152.
- [14] Pruijm M, Milani B, Burnier M. Blood oxygenation level-dependent mri to assess renal oxygenation in renal diseases: Progresses and challenges. Front Physiol 2017;7:1–7. https://doi.org/10.3389/fphys.2016.00667.
- [15] Heyman SN, Khamaisi M, Rosen S, Rosenberger C. Renal parenchymal hypoxia, hypoxia response and the progression of chronic kidney disease. Am J Nephrol 2008;28:998–1006. https://doi.org/10.1159/000146075.

Date: 29-08-2023 Protocol version: 01.01.3

[16] Inoue T, Kozawa E, Okada H, Inukai K, Watanabe S, Kikuta T, et al. Noninvasive evaluation of kidney hypoxia and fibrosis using magnetic resonance imaging. J Am Soc Nephrol 2011;22:1429–34. https://doi.org/10.1681/ASN.2010111143.

- [17] Pruijm M, Mendichovszky IA, Liss P, Van der Niepen P, Textor SC, Lerman LO, et al. Renal blood oxygenation level-dependent magnetic resonance imaging to measure renal tissue oxygenation: a statement paper and systematic review. Nephrol Dial Transplant 2018;33:ii22–8. https://doi.org/10.1093/ndt/gfy243.
- [18] Laursen JC, Søndergaard-Heinrich N, Haddock B, Rasmussen IKB, Hansen CS, Larsson HBW, et al. Kidney oxygenation, perfusion and blood flow in people with and without type 1 diabetes. Clin Kidney J 2022;15:2072–80. https://doi.org/10.1093/ckj/sfac145.
- [19] Wilcox WR, Oliveira JP, Hopkin RJ, Ortiz A, Banikazemi M, Feldt-Rasmussen U, et al. Females with Fabry disease frequently have major organ involvement: Lessons from the Fabry Registry. Mol Genet Metab 2008;93:112–28. https://doi.org/10.1016/j.ymgme.2007.09.013.
- [20] Deegan PB, Baehner AF, Barba Romero MA, Hughes DA, Kampmann C, Beck M. Natural history of Fabry disease in females in the Fabry Outcome Survey. J Med Genet 2006;43:347–52. https://doi.org/10.1136/jmg.2005.036327.
- [21] Warnock DG, Thomas CP, Vujkovac B, Campbell RC, Charrow J, Laney DA, et al. Antiproteinuric therapy and Fabry nephropathy: Factors associated with preserved kidney function during agalsidase-beta therapy. J Med Genet 2015;52:860–6. https://doi.org/10.1136/jmedgenet-2015-103471.
- [22] Hughes DA, Aguiar P, Deegan PB, Ezgu F, Frustaci A, Lidove O, et al. Early indicators of disease progression in Fabry disease that may indicate the need for disease-specific treatment initiation: Findings from the opinion-based PREDICT-FD modified Delphi consensus initiative. BMJ Open 2020;10. https://doi.org/10.1136/bmjopen-2019-035182.
- [23] Journal O, Society I. KDIGO 2012 Clinical Practice Guideline for the Evaluation and Management of Chronic Kidney Disease 2013;3.
- [24] Laursen JC, Søndergaard-Heinrich N, de Melo JML, Haddock B, Rasmussen IKB, Safavimanesh F, et al. Acute effects of dapagliflozin on renal oxygenation and perfusion in type 1 diabetes with albuminuria: A randomised, double-blind, placebo-controlled crossover trial. EClinicalMedicine 2021;37:100895. https://doi.org/10.1016/j.eclinm.2021.100895.
- [25] Appendiks 2. Retningslinjer om anvendelse af ioniserende stråling i sundhedsvidenskabelige forsøg. Den Natl Vidensk Komité 2011;2:2–4.

Date: 29-08-2023

Protocol version: 01.01.3

# Overview of Appendix

- Informed consent form
  - o Participation in study (Patient with Fabry)
  - o Participation in study (Healthy control)
  - o Biobank of future research
- Documentation of Primary
- Curriculum Vitae of Primary
- Participant information
- Information Pamphlets
  - o "Forsøgspersonens rettigheder i et sundhedsvidenskabeligt forskningsprojekt"
  - o "Dit væv, din ret"
- Questionnaires
  - o SF-36 Quality of Life questionnaire